CLINICAL TRIAL: NCT03748901
Title: A Retrospective Multicenter Analysis of PD-L1 Expression in Japanese Renal Cell Carcinoma Patients
Brief Title: PD-L1 Expression in Japanese Renal Cell Carcinoma Patients
Status: Completed | Type: Observational
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: CMA-Ate004
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Full analysis set: Patients with recurrent or metastatic RCC who have initiated first line treatment between 1 January 2010 and 31 December 2015, with representative FFPE of nephrectomy surgical specimen which are suitable for assessment of PD-L1 expression

SUMMARY:
This is a multicenter retrospective study designed to compare overall survival (OS) by PD-L1 expression status in patients with RCC who have received systemic chemotherapy for recurrent or metastatic RCC, to determine whether the prognosis is worse in PD-L1-positive than in PD-L1-negative RCC.

Total 600 RCC surgical specimens will be collected from patients who started systemic chemotherapy for recurrent or metastatic RCC between January 1, 2010 and December 31, 2015 at about 30 participating study sites in Japan.

PD-L1 expression status (IC; immune cell) on tumor-infiltrating immune cells will be evaluated by IHC, and classified by score: IC0 (PD-L1-negative) and IC1, IC2, IC3 (PD-L1-positive). Unless otherwise specified, between-group comparisons will be performed between IC0 and IC1/2/3.

ELIGIBILITY:
Inclusion Criteria:

* 1. Written informed consent for this study. In the case obtaining written informed consent is difficult due to death, change of address, and so on, the opt-out consent is accepted by giving patients or their relatives notification regarding the usage of their clinical information and surgical samples for the research.
* 2. Age at nephrectomy≧20 years
* 3.Patients with recurrent or metastatic RCC who have initiated first line treatment between 1 January 2010 and 31 December 2015, with representative FFPE of nephrectomy surgical specimen which are suitable for assessment of PD-L1 expression

Exclusion Criteria:

* 1. Malignancies other than RCC is co-existed from the time of nephrectomy and death.
* 2. Treatment with anti-CTLA-4 antibody, anti-PD-1/PD-L1 antibodies as first-line therapy for recurrent or metastatic RCC.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recurrent or metastatic RCC who have initiated first line treatment between 1 January 2010 and 31 December 2015, with representative FFPE of nephrectomy surgical specimen which are suitable for assessment of PD-L1 expression
Sampling Method: Non-Probability Sample
Enrollment: 830 (Actual)
Dates: Start 2018-12-16 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
Overall survival in PD-L1 negative (IC0) and positive (IC1/2/3) patients. | Baseline
  Overall survival is defined as the time from the initiation date of first line treatment to death due to any cause.

SECONDARY OUTCOMES:
Overall survival by PD-L1 expression status (IC0, IC1, IC2, IC3) | Baseline
  Overall survival is defined as the time from the initiation date of first line treatment to death due to any cause.
Overall survival after nephrectomy (including cytoreductive nephrectomy) | Baseline
  Overall survival is defined the time from nephrectomy (including cytoreductive nephrectomy) to death due to any cause.
Time to recurrence after radical nephrectomy | Baseline
  Time to recurrence after radical nephrectomy is the duration from the day of surgery to diagnosis of recurrent.
Treatment duration (first-line and second-line therapy) | Baseline
  Treatment duration is the duration from the day1 of systemic therapy for mRCC to the end of the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Aichi Medical University, Nagoya, Aichi-ken, Japan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (ClinicalStudyDataRequest.com). For further details on Chugai's Data Sharing Policy and how to request access to related clinical study documents, see here (www.chugai-pharm.co.jp/english/profile/rd/ctds_request.html)